CLINICAL TRIAL: NCT05275140
Title: Effectiveness of Adapted Taekwondo, Multi-component Training and Walking on Health Status in Independent Older Women: a Randomized Controlled Trial With Group and Inter-individual Analysis
Brief Title: Adapted Taekwondo on Health Status in Older Women
Acronym: TKD&Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Pablo Valdés-Badilla, Academic-Researcher at the Department of Physcial Activity Sciences, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11220035
Record Dates: First submitted 2022-01-14; First posted 2022-03-11 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Healthy People Programs
Keywords: Public health; Physical Activity; Older adults; Active aging; Combat sports.
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Physical Fitness

STUDY DESIGN:
Intervention Model Description: The study includes an experimental design (randomized controlled trial), double-blind, with repeated measures, parallel groups and a quantitative approach.
Who Masked: Participant, Outcomes Assessor
Masking Description: The assessments will be scheduled one week before and after the intervention with a team of evaluators who will not have information about the training groups, nor will the participants know their identities. That is, a double-blind shield
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group 1 (adapted taekwondo) (Experimental): The general structure of the adapted taekwondo will include a 10-min warm-up consisting of joint mobility exercises and low intensity aerobic work, then, for 40-min of the adapted taekwondo (will consist of non-contact activities, distributed in 10-min of basic postures and specific movements with the upper limbs and 20-min of lower limb movements performed individually and in pairs with and without the implementation of taekwondo. In addition, choreographies or forms (sequence of arm and leg movements that simulate an imaginary combat) specific to this modality were adapted to the characteristics of older women for 10-min; and will be developed to finish with the cool down for 10-min through dynamic and static flexibility exercises.
  Interventions: Other: Physical activity
- Experimental group 2 (multi-component training) (Active Comparator): The general structure of the multi-component training will include a 10-min warm-up consisting of joint mobility exercises and low intensity aerobic work, then, for 40-min of the multi-component training (distributed work in a circuit, which includes resistance training focused on the large muscles of the upper limbs and lower limbs combined with exercises aimed at cardiorespiratory fitness, agility and postural control, using elastic bands, poles, 2-kg medicine balls and chairs). The training volume will start (the first 4-weeks) with 3 sets of 10 repetitions per muscular exercise with a 2-min rest period between sets, performing slow movements of two seconds in concentric contraction and four seconds in eccentric contraction. Between weeks 5 to 8, the volume will increase to 4 sets of 10 repetitions per muscular exercise with 2-min of rest between sets.
  Interventions: Other: Physical activity
- Experimental group 3 (walking program) (Active Comparator): The walking program will be distributed in three weekly sessions of 45- to 60-min every other day, for 16-weeks (48 sessions). The general structure of the protocol will include a 5-min warm-up consisting of joint mobility and flexibility exercises. Next, the main part will be developed for 30- to 45-min (increased by 5-min every 4-weeks) consisting of walking on flat ground, touring the jogging circuit that the University has on campus, and ending with 5-min cool down through dynamic and static flexibility exercises.
  Interventions: Other: Physical activity
- Control group (No Intervention): The control group, the individuals will participate in the assessments (initial and final) and will be asked to maintain their usual activities. An undergraduate student (support personnel) will contact the participants by telephone (once a week) to consult them about their health status and monitor their activities. At the end of the intervention period, the control group will be invited to participate in a physical activity program that will be developed at the University based on the results of this project.

INTERVENTIONS:
Other: Physical activity — Combat sports and exercise
  Other Names: Physical fitness
  Arms: Experimental group 1 (adapted taekwondo); Experimental group 2 (multi-component training); Experimental group 3 (walking program)

SUMMARY:
The main aim of this project is to analyze and compare the effects of an adapted taekwondo program with respect to multi-component training and walking program on health status in independent older women. The study includes an experimental design (randomized controlled trial), double-blind, with repeated measures, parallel groups and a quantitative approach. The sample will be 64 women without health problems, between 60 and 65 years old and who decide to participate voluntarily. The participants will be randomized and distributed into four groups: experimental group 1 (adapted taekwondo), experimental group 2 (multi-component training), experimental group 3 (walking program) and a control group (no intervention). Assessments will consist of: systolic and diastolic blood pressure with automatic blood pressure monitor; lipid profile with the Cardiochek meter; frequency of food consumption with the modified dietary habits survey for older people; body composition by direct anthropometry and bioimpedance; cognitive status with the survey of memory, phonetic fluency and temporal-spatial orientation (in Spanish, MEFO); brain activity by means of surface electromyography; quality of life perception with the Health Survey Short Form (SF-36) version 2; physical-functional fitness with the Senior Fitness Test; handgrip strength with a hydraulic dynamometer; and postural balance with a force platform. Assessments will be performed before the 16-week intervention and after the intervention. To analyze the pre-and post-intervention results, repeated measures ANOVA will be applied for group factors (EG1 vs. EG2 vs. EG3 vs. CG) and time (pre-and post-intervention) with the Bonferroni post-hoc test; the reliability of the evaluations will be verified by means of the coefficient of intraclass correlation, and the inter-individual variability to the intervention (responders vs. non-responders) will be calculated using the technical error of measurement. The expected results indicate that adapted taekwondo produces significantly greater effects and a more favorable inter-individual response in cognitive status, brain activity, quality of life perception and postural balance compared to a multi-component training and walking program, in addition to producing similar effects at the group and inter-individual level for blood pressure, lipid profile, frequency of food consumption, body composition and physical-functional fitness in independent older women.

DETAILED DESCRIPTION:
Design The study includes an experimental design (randomized controlled trial), double-blind, with repeated measures, parallel groups and a quantitative approach. Sixty-four women over 60 years of age will be invited to participate in the study voluntarily and then be electronically randomized (https://www.randomizer.org/) and assigned to either experimental group 1 (EG1, n = 16; adapted taekwondo), experimental group 2 (EG2, n = 16; multi-component training), experimental group 3 (EG3, n = 16, walking program) or the control group (CG, n = 16; no intervention).

Sample The sample calculation indicates that the ideal number of participants per group is 16. According to previous research, for this calculation, an average difference of 3.46 repetitions (chair stand test) was used as the minimum difference required for substantial clinical relevance, with a standard deviation of 3.38 repetitions, considering an alpha level of 0.05 with 90% power and an expected loss of 15%. The inclusion criteria for the sample will be: i) older women aged between 60 and 65 years old; ii) presenting the ability to understand and follow instructions in a contextualized way through simple commands; iii) independent, that is, have a score equal to or greater than 43 points in the Preventive Medicine Exam for the Older People (in Spanish, EMPAM) of the Ministry of Health (31); and iv) complying with at least 85% attendance at the sessions scheduled for interventions. Regarding the exclusion criteria, the following will be considered: i) having any disabling disease; ii) those women who have musculoskeletal injuries or who are undergoing physical rehabilitation treatment that prevents their normal physical performance; and iii) those who have permanent or temporary contraindications to perform PA.

All participants will be informed of the scope of the research and will sign an informed consent that authorizes the use of the information for scientific purposes. In addition, the research protocol will follow the CONSORT guidelines, will be reviewed by the Scientific Ethics Committee of the Universidad Católica del Maule and will be developed following what is stated in the Declaration of Helsinki for work with human beings.

Before starting the intervention, during the last week of July 2022 (for one week), older women will be evaluated in the variables considered for the research, later, from the first week of August to the last week of November 2022 (16 weeks) will participate in designated training programs. After the intervention (first week of December 2022), for one week, the older women will undergo the same initial assessments.

ELIGIBILITY:
Inclusion Criteria:

* Older women aged between 60 and 65 years old.
* Presenting the ability to understand and follow instructions in a contextualized way through simple commands.
* Independent, that is, have a score equal to or greater than 43 points in the Preventive Medicine Exam for the Older People (in Spanish, EMPAM) of the Ministry of Health (31).
* Complying with at least 85% attendance at the sessions scheduled for interventions.

Exclusion Criteria:

* Having any disabling disease.
* Those women who have musculoskeletal injuries or who are undergoing physical rehabilitation treatment that prevents their normal physical performance.
* Those who have permanent or temporary contraindications to perform physical activity.

Ages: 60 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Blood Pressure at 16 weeks | 2 weeks
  The systolic and diastolic blood pressure will be obtained with an automatic pressure monitor (08A, CONTEC, Germany). The participants will be evaluated considering at least 10-min of previous rest in a sitting position, with the back and arms supported and the legs without crossing, emptying the urinary bladder if necessary. In addition, women will be asked not to do exercise, smoke, drink alcohol or coffee at least 30-min before the measurements. The first assessment will be taken in both arms to identify the arm with the highest blood pressure, and then two assessments will be taken in the arm with the highest blood pressure (usually the dominant) adding a third assessment if the difference between the measurements is greater than 5 mmHg.
Change from Lipid Profile at 16 weeks | 2 weeks
  This will be determined in a fasting condition of at least 12-h; the extraction of 5 ml of capillary blood will be carried out by a nurse considering the necessary safeguards in the Human Performance Laboratory with the use of a meter (Cardiochek PA, USA) to determine total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, cholesterol without HDL, and total cholesterol/HDL cholesterol ratio.
Change from Frequency of Food Consumption at 16 weeks | 2 weeks
  The aim of the survey is to measure the eating habits of older people and is made up of two areas of self-application. The first is composed of 12 items with a minimum score of 1 and a maximum of 5 per question (Likert scale), which indicates the frequency of healthy habits, such as the frequency of consumption of recommended food groups, ranging from not consuming (1 point) up to the suggested day/week servings (5 points), with a score of the responses that varies from 12 to 60 points (higher value, better eating habits). The second area consists of 7 items, foods or food groups identified as promoters of chronic non-communicable diseases (sugary drinks, alcohol, fried foods, fast food, sweet snacks, coffee), and a negative eating habit is added, such as adding salt to meals without tasting them; reaching a value that ranges from 7 to 33 points (higher values indicate worse eating habits).
Change from Anthropometric measurements at 16 weeks | 2 weeks
  The following anthropometric measurements will be obtained: i) body weight in kg with a digital scale (Seca 769, Germany; Accuracy of 0.1 kg); ii) bipedal height in cm with a stadiometer (Seca 220, Germany; Accuracy of 0.1 cm). Weight and height will be combined to report BMI in kg/m^2.
Change from Body Composition (muscle mass) at 16 weeks | 2 weeks
  The following body composition (muscle mass) will be obtained: i) diameters (biacromial, transverse thorax, anteroposterior thorax, bi-iliocrestid, humeral, femoral) in cm with an anthropometer (Rosscraft Campbell 20; Accuracy of 0.1 mm); ii) perimeters (head, arm relaxed, arm flexed in tension, forearm maximum, mesosternal thorax, minimum waist, maximum hip, maximum thigh, medial thigh, maximum calf) in cm using an inextensible measuring tape (Seca 201, Germany); and iii) skinfolds (tricipital, subscapular, supraspinal, abdominal, medial thigh, calf) in mm with a caliper (Harpenden, England; Accuracy of 0.2 mm.
Change from Body Composition (fat mass) at 16 weeks | 2 weeks
  The following body composition (fat mass) will be obtained: i) diameters (biacromial, transverse thorax, anteroposterior thorax, bi-iliocrestid, humeral, femoral) in cm with an anthropometer (Rosscraft Campbell 20; Accuracy of 0.1 mm); ii) perimeters (head, arm relaxed, arm flexed in tension, forearm maximum, mesosternal thorax, minimum waist, maximum hip, maximum thigh, medial thigh, maximum calf) in cm using an inextensible measuring tape (Seca 201, Germany); and iii) skinfolds (tricipital, subscapular, supraspinal, abdominal, medial thigh, calf) in mm with a caliper (Harpenden, England; Accuracy of 0.2 mm.
Change from Body Composition (fat mass) by bioimpedance at 16 weeks | 2 weeks
  The following body composition (bioimpedance), the percentage of fat mass will be obtained using eight electrode tetrapolar bioimpedance (InBody 570®, Body Composition Analyzers, South Korea).
Change from Body Composition (fat-free mass) by bioimpedance at 16 weeks | 2 weeks
  The following body composition (bioimpedance), the percentage of fat-free mass will be obtained using eight electrode tetrapolar bioimpedance (InBody 570®, Body Composition Analyzers, South Korea).
Change from Cognitive Status at 16 weeks | 2 weeks
  This will be evaluated using the memory, phonetic fluency and temporal-spatial orientation survey (in Spanish, MEFO) (34), which aims to determine the level of cognitive impairment in older people. This survey classifies the participants into three levels: without cognitive impairment, with mild cognitive impairment, or with cognitive impairment. The advantage of the MEFO is that the level of schooling does not have an influence; its application is simple and brief (34). The MEFO assesses deferred free recall, phonetic fluency with the letter P, and temporal-spatial orientation; furthermore, it has high sensitivity in the fields described and is validated for use with older people in Chile (34).
Change from Brain Activity at 16 weeks | 2 weeks
  This will be analyzed through a 64+8 channel surface electromyography system (active-Two from BioSemi, The Netherlands) using a mapping task and a reaction time task, with the aim of measuring spatial and visual-abilities motor skills, in addition to the planning index of the participants, following previous recommendations (35).
Change from Quality of Life Perception at 16 weeks | 2 weeks
  This will be obtained using the Health Survey Short Form (SF-36) version 2, which measures the attributes of eight health dimensions: physical function, physical role, body pain, general health, vitality, social function, emotional role and mental health (36). Each dimension is made up of a series of questions that together give a scale ranging from 0 (the worst health status for that dimension) to 100 (the best health status) (36).
Change from Physical-Functional Fitness (strenght of the lower body) at 16 weeks | 2 weeks
  This will be evaluated with the Senior Fitness Test, which allows evaluation of great reliability and easy application (37). The chair stand test to assess the strength of the lower body, counting the number of repetitions made in 30s.
Change from Physical-Functional Fitness (strenght on the upper body) at 16 weeks | 2 weeks
  This will be evaluated with the Senior Fitness Test, which allows evaluation of great reliability and easy application (37). The arm curl test to assess the strength on the upper body, using a 3lb (women) and 5lb (men) dumbbell, counting the number of repetitions made in 30s.
Change from Physical-Functional Fitness (aerobic fitness) at 16 weeks | 2 weeks
  This will be evaluated with the Senior Fitness Test, which allows evaluation of great reliability and easy application (37). The 2-minute step to assess aerobic fitness, recording the number of knee elevations.
Change from Physical-Functional Fitness (flexibility of the lower-body) at 16 weeks | 2 weeks
  This will be evaluated with the Senior Fitness Test, which allows evaluation of great reliability and easy application (37). The chair sit-&-reach test to assess the flexibility of the lower-body, measured in cm.
Change from Physical-Functional Fitness (flexibility on the upper-body) at 16 weeks | 2 weeks
  This will be evaluated with the Senior Fitness Test, which allows evaluation of great reliability and easy application (37). The back scratch test to assess flexibility on the upper-body, measured in cm.
Change from Physical-Functional Fitness (agility and dynamic balance) at 16 weeks | 2 weeks
  This will be evaluated with the Senior Fitness Test, which allows evaluation of great reliability and easy application (37). The timed up-and-go test to assess agility and dynamic balance, surrounding a cone at 8ft (2.44m) and recording time in seconds.
Change from Handgrip Strength at 16 weeks | 2 weeks
  The handgrip strength will be measured with a hydraulic dynamometer (Camry, model EH101, China)
Change from Postural Balance at 16 weeks | 2 weeks
  The postural balance will be obtained with a force platform (ArtOficio Ltda., Chile).

SECONDARY OUTCOMES:
Sociodemographic Assessments | 1 week
  Age (years), academic level (primary, secondary, bachelor, master, PhD), civil status (married, separated, widow, single, others).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Valdés-Badilla, PhD, Principal Investigator — Universidad Católica del Maule
Locations (1):
- Poliderportivo San Clemente, San Clemente, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared. We will only disseminate the results of the study through scientific papers and presentations at scientific congresses

REFERENCES:
- [Background] Yerrakalva D, Yerrakalva D, Hajna S, Griffin S. Effects of Mobile Health App Interventions on Sedentary Time, Physical Activity, and Fitness in Older Adults: Systematic Review and Meta-Analysis. J Med Internet Res. 2019 Nov 28;21(11):e14343. doi: 10.2196/14343. PMID 31778121
- [Background] Zubala A, MacGillivray S, Frost H, Kroll T, Skelton DA, Gavine A, Gray NM, Toma M, Morris J. Promotion of physical activity interventions for community dwelling older adults: A systematic review of reviews. PLoS One. 2017 Jul 10;12(7):e0180902. doi: 10.1371/journal.pone.0180902. eCollection 2017. PMID 28700754
- [Background] Grande GD, Oliveira CB, Morelhao PK, Sherrington C, Tiedemann A, Pinto RZ, Franco MR. Interventions Promoting Physical Activity Among Older Adults: A Systematic Review and Meta-Analysis. Gerontologist. 2020 Nov 23;60(8):583-599. doi: 10.1093/geront/gnz167. PMID 31868213
- [Background] Fragala MS, Cadore EL, Dorgo S, Izquierdo M, Kraemer WJ, Peterson MD, Ryan ED. Resistance Training for Older Adults: Position Statement From the National Strength and Conditioning Association. J Strength Cond Res. 2019 Aug;33(8):2019-2052. doi: 10.1519/JSC.0000000000003230. PMID 31343601
- [Background] Chang YK, Pan CY, Chen FT, Tsai CL, Huang CC. Effect of resistance-exercise training on cognitive function in healthy older adults: a review. J Aging Phys Act. 2012 Oct;20(4):497-517. doi: 10.1123/japa.20.4.497. Epub 2011 Dec 20. PMID 22186664
- [Background] Valdes-Badilla PA, Gutierrez-Garcia C, Perez-Gutierrez M, Vargas-Vitoria R, Lopez-Fuenzalida A. Effects of Physical Activity Governmental Programs on Health Status in Independent Older Adults: A Systematic Review. J Aging Phys Act. 2019 Apr 1;27(2):265-275. doi: 10.1123/japa.2017-0396. Epub 2018 Nov 13. PMID 29989461
- [Background] McAuley PA, Artero EG, Sui X, Lee DC, Church TS, Lavie CJ, Myers JN, Espana-Romero V, Blair SN. The obesity paradox, cardiorespiratory fitness, and coronary heart disease. Mayo Clin Proc. 2012 May;87(5):443-51. doi: 10.1016/j.mayocp.2012.01.013. Epub 2012 Apr 12. PMID 22503065
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Reis RS, Salvo D, Ogilvie D, Lambert EV, Goenka S, Brownson RC; Lancet Physical Activity Series 2 Executive Committee. Scaling up physical activity interventions worldwide: stepping up to larger and smarter approaches to get people moving. Lancet. 2016 Sep 24;388(10051):1337-48. doi: 10.1016/S0140-6736(16)30728-0. Epub 2016 Jul 28. PMID 27475273
- [Background] Galloza J, Castillo B, Micheo W. Benefits of Exercise in the Older Population. Phys Med Rehabil Clin N Am. 2017 Nov;28(4):659-669. doi: 10.1016/j.pmr.2017.06.001. PMID 29031333
- [Background] Ramirez-Campillo R, Alvarez C, Garcia-Hermoso A, Celis-Morales C, Ramirez-Velez R, Gentil P, Izquierdo M. High-speed resistance training in elderly women: Effects of cluster training sets on functional performance and quality of life. Exp Gerontol. 2018 Sep;110:216-222. doi: 10.1016/j.exger.2018.06.014. Epub 2018 Jun 15. PMID 29909049
- [Background] Martinez-Velilla N, Casas-Herrero A, Zambom-Ferraresi F, Saez de Asteasu ML, Lucia A, Galbete A, Garcia-Baztan A, Alonso-Renedo J, Gonzalez-Glaria B, Gonzalo-Lazaro M, Apezteguia Iraizoz I, Gutierrez-Valencia M, Rodriguez-Manas L, Izquierdo M. Effect of Exercise Intervention on Functional Decline in Very Elderly Patients During Acute Hospitalization: A Randomized Clinical Trial. JAMA Intern Med. 2019 Jan 1;179(1):28-36. doi: 10.1001/jamainternmed.2018.4869. PMID 30419096
- [Background] Das Gupta S, Bobbert MF, Kistemaker DA. The Metabolic Cost of Walking in healthy young and older adults - A Systematic Review and Meta Analysis. Sci Rep. 2019 Jul 10;9(1):9956. doi: 10.1038/s41598-019-45602-4. PMID 31292471
- [Background] Fonseca Alves DJ, Bartholomeu-Neto J, Junior ER, Ribeiro Zarricueta BS, Nobrega OT, Cordova C. Walking Speed, Risk Factors, and Cardiovascular Events in Older Adults-Systematic Review. J Strength Cond Res. 2017 Nov;31(11):3235-3244. doi: 10.1519/JSC.0000000000002182. PMID 29065080
- [Background] Chen YW, Hunt MA, Campbell KL, Peill K, Reid WD. The effect of Tai Chi on four chronic conditions-cancer, osteoarthritis, heart failure and chronic obstructive pulmonary disease: a systematic review and meta-analyses. Br J Sports Med. 2016 Apr;50(7):397-407. doi: 10.1136/bjsports-2014-094388. Epub 2015 Sep 17. PMID 26383108
- [Background] Cho SY, Roh HT. Taekwondo Enhances Cognitive Function as a Result of Increased Neurotrophic Growth Factors in Elderly Women. Int J Environ Res Public Health. 2019 Mar 18;16(6):962. doi: 10.3390/ijerph16060962. PMID 30889827
- [Background] Yu AP, Tam BT, Lai CW, Yu DS, Woo J, Chung KF, Hui SS, Liu JY, Wei GX, Siu PM. Revealing the Neural Mechanisms Underlying the Beneficial Effects of Tai Chi: A Neuroimaging Perspective. Am J Chin Med. 2018;46(2):231-259. doi: 10.1142/S0192415X18500131. PMID 29542330
- [Background] Ciaccioni S, Capranica L, Forte R, Chaabene H, Pesce C, Condello G. Effects of a Judo Training on Functional Fitness, Anthropometric, and Psychological Variables in Old Novice Practitioners. J Aging Phys Act. 2019 May 31;27(4):831-842. doi: 10.1123/japa.2018-0341. Online ahead of print. PMID 31034297
- [Background] Bromley SJ, Drew MK, Talpey S, McIntosh AS, Finch CF. A systematic review of prospective epidemiological research into injury and illness in Olympic combat sport. Br J Sports Med. 2018 Jan;52(1):8-16. doi: 10.1136/bjsports-2016-097313. Epub 2017 Sep 27. PMID 28954799
- [Background] Lee SH, Scott SD, Pekas EJ, Lee S, Lee SH, Park SY. Taekwondo training reduces blood catecholamine levels and arterial stiffness in postmenopausal women with stage-2 hypertension: randomized clinical trial. Clin Exp Hypertens. 2019;41(7):675-681. doi: 10.1080/10641963.2018.1539093. Epub 2018 Nov 2. PMID 30388905
- [Background] Valdes-Badilla PA, Godoy-Cumillaf A, Ortega-Spuler J, Diaz-Aravena D, Castro-Garrido N, Sandoval-Munoz L, Herrera-Valenzuela T, Lopez-Fuenzalida A, Vargas-Vitoria R, Duran-Aguero S. [Relationship between anthropometric health indexes with food consumption in physically active elderly]. Nutr Hosp. 2017 Oct 24;34(5):1073-1079. doi: 10.20960/nh.1012. Spanish. PMID 29130704
- [Background] Basso D, Saracini C. Differential involvement of left and right frontoparietal areas in visuospatial planning: An rTMS study. Neuropsychologia. 2020 Jan;136:107260. doi: 10.1016/j.neuropsychologia.2019.107260. Epub 2019 Nov 14. PMID 31734226
- [Background] Vilagut G, Ferrer M, Rajmil L, Rebollo P, Permanyer-Miralda G, Quintana JM, Santed R, Valderas JM, Ribera A, Domingo-Salvany A, Alonso J. [The Spanish version of the Short Form 36 Health Survey: a decade of experience and new developments]. Gac Sanit. 2005 Mar-Apr;19(2):135-50. doi: 10.1157/13074369. Spanish. PMID 15860162
- [Background] Valdes-Badilla P, Herrera-Valenzuela T, Ramirez-Campillo R, Aedo-Munoz E, Baez-San Martin E, Ojeda-Aravena A, Branco BHM. Effects of Olympic Combat Sports on Older Adults' Health Status: A Systematic Review. Int J Environ Res Public Health. 2021 Jul 10;18(14):7381. doi: 10.3390/ijerph18147381. PMID 34299833
- See also: Ministerio de Salud. Programa Más Adultos Mayores Autovalentes — http://bit.ly/3hoPqQ8
- See also: Ministerio de Salud. Encuesta Nacional de Salud 2016-2017 — https://www.minsal.cl/wp-content/uploads/2017/11/ENS-2016-17_PRIMEROS-RESULTADOS.pdf
- See also: Ministerio del Deporte. Encuesta Nacional de Hábitos de Actividad Física y Deporte 2018 en Población de 18 años y más. — http://www.mindep.cl/secciones/151
- See also: Ministerio de Salud. Manual de Aplicación del Examen de Medicina Preventiva del Adulto Mayor — http://bit.ly/2UzMh68
- See also: International standards for anthropometric assessment. Wellington: ISAK, 2012. — http://repository.openpolytechnic.ac.nz/handle/11072/1510